CLINICAL TRIAL: NCT05114785
Title: PReserved Ejection Fraction Evaluation and Recognition by Cardiac Magnetic Resonance
Brief Title: Heart Failure With Preserved Ejection Fraction: Evaluation and Recognition by CMR
Acronym: PREFER-CMR
Status: Not yet recruiting | Type: Observational
Sponsor: University of East Anglia (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 301141
Record Dates: First submitted 2021-09-28; First posted 2021-11-10 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Heart Diseases
Keywords: Heart failure; hemodynamics; magnetic resonance imaging
MeSH Terms: conditions — Heart Diseases; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFpEF group: Suspected HFpEF group: 80 patients will be recruited with history of dyspnoea, LV ejection fraction ≥ 50%, raised NTproBNP
  Interventions: Diagnostic Test: Multi Parametric Cardiac Magnetic Resonance
- Control group: 20 patients with suspected CAD but with no dyspnoea and normal echocardiogram.
  Interventions: Diagnostic Test: Multi Parametric Cardiac Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Multi Parametric Cardiac Magnetic Resonance — Research based Cardiac MRI evaluation to determine cardiovascular haemodynamics

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is a common and growing condition with a poor prognosis but the pathophysiology and management are still being investigated. The PREFER-CMR project aims to evaluate and validate the application of novel 4D cardiac magnetic resonance flow dynamic methods to measure left ventricular pressures and validate these measurements with direct pressure measurement by coronary angiography. This is a prospective observational study of patients with HFpEF undergoing clinical evaluation with coronary angiography who will also undergo contemporaneous cardiac MRI. The primary outcome will be the level of agreement between the two methods using angiography as the reference method.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is prevalent, increasing in incidence and has a poor prognosis. Accurate left ventricular (LV) haemodynamic assessment is needed to diagnose and manage patients with HFpEF. The reference method for assessment is an invasive study using catheters to measure intra-ventricular pressure but this is rarely done due to its invasive nature, high procedural costs and lack of expertise, despite the fact that haemodynamic guided therapy is associated with reduced re-hospitalisation and mortality. Non-invasive methods of LV haemodynamic assessment are inaccurate. The Investigators have developed an accurate four-dimensional flow cardiac magnetic resonance (4D flow CMR) protocol which is non-invasive and addresses the issues with existing practices to evaluate HFpEF. This observational-analytical study aims to assess the utility of a non-invasive 4D flow CMR protocol for haemodynamic assessment of HFpEF, to generate clinical data to support future clinical trials, clinical translation and patient benefit. This research study will involve generating a precise haemodynamic model using invasive and non-invasive data of prospectively recruited patients. This model will be also optimised in clinical patients with arrhythmias. Also, observational data will be collected to test the model's prognostic value.

ELIGIBILITY:
Inclusion Criteria:

1. Adults: age≥18 years.
2. Typical HF symptoms (NYHA stage>I) within the last six months.
3. Raised NTproBNP (>400 pg/ml)
4. EF>50 % with the absence of structural heart disease on TTE (except left ventricular hypertrophy or left atrial enlargement).

Exclusion Criteria:

1. Patients unable/unwilling to provide informed consent.
2. Bodyweight>120 kg or inability to lie flat/still.
3. Contraindication for invasive workup (allergy to contrast, severe renal insufficiency with estimated glomerular filtration rate (eGRF)<30 ml/min).
4. Contraindications for a contrast-enhanced CMR study (allergy to contrast, incompatible devices or implants, severe claustrophobia).
5. Previous medical history of EF <50%
6. Pregnancy

The extended observational arm of the study will have wider eligibility criteria

- Patients undergoing cardiac MRI for clinical indications irrespective of EF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Suspected heart failure patients
  * Suspected coronary artery disease patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Left ventricular pressure measured by invasive angiography (reference method) and modelled by cardiovascular magnetic resonance imaging | 30 days
  Agreement of invasively measured left ventricular pressure in millimeters of mercury (mmHg) by invasive angiography to non-invasively modelled left ventricular pressure by cardiac magnetic resonance imaging. The agreement will be tested by Bland-Altman plots..

SECONDARY OUTCOMES:
Prognostic relevance of left ventricular pressures measured by cardiac MRI | Ten years
  Is cardiovascular magnetic resonance modelled left ventricular pressure in millimeters of mercury (mmHg) associated with MACE events including re-hospitalization, stroke, myocardial infarction and death. Association between pressure measurements and MACE will be tested by Cox proportional hazards regression and Kaplan-Meier survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Pankaj Garg, MD, Principal Investigator — University of East Anglia

IPD SHARING:
Plan to Share IPD: Yes
The dataset of this study are available at the discretion of the Principal Investigator on reasonable request.

REFERENCES:
- [Derived] Bana A, Li R, Mehmood Z, Rogers C, Grafton-Clarke C, Bali T, Hall D, Jamil M, Ramachenderam L, Dudhiya U, Spohr H, Underwood V, Girling R, Kasmai B, Nair S, Matthews G, Garg P. Does CMR improve aetiological sub-phenotyping beyond echocardiography in patients with elevated LV filling pressure? A prospective registry study (PREFER-CMR). BMJ Open. 2026 Jan 14;16(1):e102836. doi: 10.1136/bmjopen-2025-102836. PMID 41535077
- [Derived] Grafton-Clarke C, Assadi H, Li R, Mehmood Z, Hall R, Matthews G, Tsampasian V, Alabed S, Kasmai B, Staff L, Curtin J, Yashoda GK, Sun J, Nair S, Hewson D, Thampi K, Broncano J, Ricci F, Swoboda P, Swift AJ, Vassiliou VS, Geest RJV, Garg P. Four-dimensional flow provides incremental diagnostic value over echocardiography in aortic stenosis. Open Heart. 2025 May 7;12(1):e003081. doi: 10.1136/openhrt-2024-003081. PMID 40340893
- [Derived] Assadi HS, Zhao X, Matthews G, Li R, Broncano Cabrero J, Kasmai B, Alabed S, Royuela Del Val J, Spohr H, Gurung-Koney Y, Aung N, Nair S, Swift AJ, Vassiliou VS, Zhong L, Al-Mohammad A, van der Geest RJ, Swoboda PP, Plein S, Garg P. Cardiovascular magnetic resonance imaging markers of ageing: a multi-centre, cross-sectional cohort study. Eur Heart J Open. 2025 May 2;5(3):oeaf032. doi: 10.1093/ehjopen/oeaf032. eCollection 2025 May. PMID 40322642
- [Derived] Assadi H, Sawh C, Spohr H, Nelthorpe F, Nair S, Hughes M, Ashman D, Ryding A, Matthews G, Li R, Grafton-Clarke C, Mehmood Z, Al-Mohammad A, Kasmai B, Vassiliou VS, Garg P. Clinical relevance of aortic conduit and reservoir function. Open Heart. 2024 Aug 19;11(2):e002713. doi: 10.1136/openhrt-2024-002713. PMID 39160086
- [Derived] Assadi H, Alabed S, Li R, Matthews G, Karunasaagarar K, Kasmai B, Nair S, Mehmood Z, Grafton-Clarke C, Swoboda PP, Swift AJ, Greenwood JP, Vassiliou VS, Plein S, van der Geest RJ, Garg P. Development and validation of AI-derived segmentation of four-chamber cine cardiac magnetic resonance. Eur Radiol Exp. 2024 Jul 12;8(1):77. doi: 10.1186/s41747-024-00477-7. PMID 38992116
- [Derived] Mehmood Z, Assadi H, Grafton-Clarke C, Li R, Matthews G, Alabed S, Girling R, Underwood V, Kasmai B, Zhao X, Ricci F, Zhong L, Aung N, Petersen SE, Swift AJ, Vassiliou VS, Cavalcante J, Geest RJV, Garg P. Validation of 2D flow MRI for helical and vortical flows. Open Heart. 2024 Mar 8;11(1):e002451. doi: 10.1136/openhrt-2023-002451. PMID 38458769